CLINICAL TRIAL: NCT02869854
Title: Increased Adherence to Physical Activity on Prescription (PAP) Through Mindfulness- A Pilot Study.
Brief Title: Increased Physical Activity Through Mindfulness
Acronym: FAR-MIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pny1
Record Dates: First submitted 2016-08-08; First posted 2016-08-17 (Estimated); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-02

CONDITIONS: Physical Activity; Life Style; Mindfulness
MeSH Terms: conditions — Motor Activity | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PAP only (Active Comparator): This group will follow the referral scheme for three months, and after this period they will leave new blood samples and answer surveys. They will get a new PAP with follow up after another 3 months.
  Interventions: Behavioral: PAP
- Mindfulness only (Active Comparator): Mindfulness. This group will receive a group course in mindfulness during 8 weeks once a week, and with 20 minutes of daily personal training. Three and six months after inclusion they will answer a new set of surveys and fasting blood samples.
  Interventions: Behavioral: Mindfulness
- Combination of the two groups (Experimental): Mindfulness and physical activity prescription. This group will get a combination of the two other groups. PAP will be prescribed during the first meeting and another one after 3 months. During the first 8 weeks once a week they will participate in a mindfulness training group and also preform 20 minutes of daily training. The same surveys as the other groups and fasting blood samples
  Interventions: Behavioral: Mindfulness; Behavioral: PAP

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness course during 8 weeks with 20 minutes mindfulness exercise each day
  Arms: Combination of the two groups; Mindfulness only
Behavioral: PAP — Physical Activity on Prescription, after 3 months a new prescription
  Arms: Combination of the two groups; PAP only

SUMMARY:
In a pilot study, 90 physically inactive patients will be opportunistically and consecutively recruited and randomized to three intervention groups: mindfulness training, Physical Activity on Prescription (PAP) or only PAP. Follow-up will be done at baseline, three and six months with questionnaires, accelerometers and analysis of traditional risk factors to evaluate whether mindfulness may increase physical activity and decrease physical inactivity.

DETAILED DESCRIPTION:
All patients between 40 and 65 years of age who fulfil the inclusion criteria will be asked to participate in the study. Posters with information about the study will be put in the waiting room and in other strategic places. Patients who accept to participate will get written and oral information; they will sign an informed consent after the information. The patients will estimate their level of physical activity in minutes per week to control inclusion criteria. The patients will return in the morning for fasting blood samples and get an accelerometer attached to them to wear for 7 days. During this time, randomization will be performed. They will also get to answer a couple of different surveys. The results from the surveys and blood samples will be the study baseline.

All patients with abnormal test results will follow a specific flow diagram for the usual care.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 40-65 years of age, with insufficient physical activity ( <150 minutes of moderate-intensity physical activity throughout the week, or < 75 minutes of vigorous-intensity physical activity throughout the week, or an equivalent combination of moderate- and vigorous-intensity activity.)

Exclusion Criteria:

* Dementia, severe mental disorder,newly diagnosed untreated unstable angina pectoris,myocardial infarction within 6 weeks prior to study entry. Individuals who do not master the Swedish language in speech and writing will be excluded.The patients who have abnormal values according to guidelines that require contact with a physician on the same day or week will also be excluded

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Zöller, Docent, Principal Investigator — Lunds University
Locations (1):
- Lunds Unniversitet, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nymberg P, Ekvall Hansson E, Stenman E, Calling S, Sundquist K, Sundquist J, Zoller B. Pilot study on increased adherence to physical activity on prescription (PAP) through mindfulness: study protocol. Trials. 2018 Oct 17;19(1):563. doi: 10.1186/s13063-018-2932-9. PMID 30333052
- [Derived] Nymberg P, Calling S, Stenman E, Palmer K, Hansson EE, Sundquist K, Sundquist J, Zoller B. Effect of mindfulness on physical activity in primary healthcare patients: a randomised controlled trial pilot study. Pilot Feasibility Stud. 2021 Mar 17;7(1):70. doi: 10.1186/s40814-021-00810-6. PMID 33731219

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PAP Only | Mindfulness Only | Combination of the Two Groups
Started | 29 | 30 | 29
Completed | 16 | 19 | 19
Not Completed | 13 | 11 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PAP Only | Mindfulness Only | Combination of the Two Groups | Total
Number analyzed (Participants) | 29 | 30 | 29 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 30 | 29 | 88
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 54 [42 to 65] | 53 [41 to 65] | 54 [43 to 64] | 54 [41 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 20 | 64
  Male | 7 | 8 | 9 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 29 | 30 | 29 | 88

OUTCOME MEASURES:

1. Primary Outcome: Difference in Percentage of Time Spent Per Physical Activity Level Per Week of Time, Between the Three Different Groups Measured by Activity Monitor Actigraph (GT3X)
Description: Each individual will wear an activity monitor for 7 days. This will be done at baseline and after 6 months. The difference in the time of physical activity level was measured in minutes of activity during a week and then divided into percentages of sedentary time, light physical activity time and moderate to vigourous physical activity time, measured by activity monitor Actigraph (GT3X). In the analysis
Time Frame: Baseline ,6 months.
Population: Baseline and 6 months follow-up after inclusion. Change in percentage of sedentary time and time in different intensity of physical activity per valid day and averaged over the number of valid days, activity monitor measured
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | PAP Only | Mindfulness Only | Combination of the Two Groups
Number analyzed (Participants) | 29 | 30 | 29
percentage of time
  Baseline:Percent of time in sedentary time | 66.2 (6.7) | 65.5 (9.2) | 66.7 (8.8)
  Baseline:Percent of time in LIPA | 30.9 (6.2) | 31.7 (8.2) | 30.3 (8.0)
  Baseline:Percent of time in MVPA | 2.6 (0.18) | 2.3 (0.02) | 2.4 (0.02)
  6 months:Percent of time in sedentary time: number analyzed (Participants) | 22 | 24 | 26
  6 months:Percent of time in sedentary time | 65.0 (6.8) | 65.9 (9.4) | 64.0 (9.1)
  6 months Percent of LIPA: number analyzed (Participants) | 22 | 24 | 26
  6 months Percent of LIPA | 32.0 (5.8) | 31.6 (9.0) | 32.8 (8.9)
  6 months: Percent of MVPA: number analyzed (Participants) | 22 | 24 | 26
  6 months: Percent of MVPA | 2.6 (0.02) | 1.9 (0.02) | 2.7 (0.02)

2. Secondary Outcome: Difference Between the Three Groups in Revised Assessment of Their Self-rated Health
Description: assessment based on terms of perceived health with five alternative answers, a higher score incdicates a better outcome
  1. very poor
  2. poor
  3. fair
  4. good
  5. very good
Time Frame: base-line ,3 months, 6 months
Population: The number decreases during the study due to dropout, lost to follow-up.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | PAP Only | Mindfulness Only | Combination of the Two Groups
Number analyzed (Participants) | 29 | 30 | 29
score on a scale
  Baseline | 3 [1 to 4] | 3 [2 to 5] | 3 [2 to 5]
  3 months: number analyzed (Participants) | 22 | 24 | 26
  3 months | 3 [1 to 4] | 3 [2 to 5] | 4 [2 to 5]
  6 months: number analyzed (Participants) | 22 | 24 | 24
  6 months | 4 [1 to 4] | 4 [2 to 5] | 4 [2 to 5]

3. Secondary Outcome: Difference Between Groups in the Amount of Self-perceived Sleep Problems
Description: Insomnia Severity Index(ISI); is a self-report questionnaire measuring insomnia symptoms to evaluate the degree of insomnia. The scale consists of seven questions that evaluate Sleep mode, sleep during the night, waking up early, the feeling of being rested, how sleeping problems affect daily life, and how sleep patterns concern the individual. The higher the score, the better the outcome. Minimun score = 0, Maximum score = 28
Time Frame: Baseline, 3 months, 6 months
Population: decreasing numbers due to drop-out
Measure: Median (Full Range); unit: score on a scale
Arm/Group | PAP Only | Mindfulness Only | Combination of the Two Groups
Number analyzed (Participants) | 29 | 30 | 29
score on a scale
  Insomnia Severity Index baseline | 8 [0 to 24] | 11 [0 to 27] | 10 [0 to 21]
  Insomnia Severity Index 3 months: number analyzed (Participants) | 22 | 24 | 26
  Insomnia Severity Index 3 months | 7 [0 to 20] | 11 [0 to 27] | 9 [0 to 27]
  Insomnia Severity Index 6 months: number analyzed (Participants) | 22 | 24 | 24
  Insomnia Severity Index 6 months | 6 [0 to 18] | 13 [0 to 25] | 9 [0 to 18]

ADVERSE EVENTS:
Time Frame: baseline, 3 months, 6 months
Description: no adverse events appeared
Arm/Group | PAP Only | Mindfulness Only | Combination of the Two Groups
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29 | 0/27
Other Adverse Events (participants affected / at risk) | 0/28 | 0/29 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2016-04-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT02869854/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT02869854/SAP_001.pdf
  • Informed Consent Form (2016-04-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT02869854/ICF_002.pdf